CLINICAL TRIAL: NCT01652196
Title: A Phase II Study of the Combination of Aflibercept (VEGF-Trap) Plus Modified FOLFOX 6 in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Aflibercept and FOLFOX6 Treatment for Previously Untreated Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Hays (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, John Hays, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU 11182; NCI-2012-01167 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IV Colon Cancer; Stage IV Rectal Cancer
Keywords: colorectal cancer; rectal cancer; FOLFOX; Aflibercept
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — aflibercept; Oxaliplatin; Leucovorin; Fluorouracil; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aflibercept (combination chemotherapy) (Experimental): Patients receive aflibercept and fluorouracil and then continuously over 46 hours on days 1 and 15.If leucovorin is not available due to drug shortages the regimen should be administered with the leucovorin omitted. Correlative Studies are required to be available before enrolling on the study. A fresh biopsy is only required if there is insufficient material for analysis. Repeat tumor biopsies after 8 weeks of therapy are optional and will only be performed at the Ohio State University Medical Center.DCE MRI (dynamic contrast-enhanced magnetic resonance imaging)images at weeks 0, and after 8 weeks +/- 1 week of treatment(after Cycle 2). 18FDG-PET is a functional imaging technique that relies on tumor uptake of radiolabeled tracer 18 fluorodeoxyglucose (18FDG).FDG-PET is a widely-used imaging modality in the detection and monitoring of a variety of metastatic cancers,including colorectal cancer (99-102).
  Interventions: Biological: aflibercept; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil; Other: Correlative Studies; Procedure: DCE MRI; Radiation: f18FDG-PET; Procedure: PET (positron emission tomography)

INTERVENTIONS:
Biological: aflibercept — 4 mg/kg as a 1-hour IV(intervenous) infusion
  Other Names: vascular endothelial growth factor trap; VEGF Trap; VEGF Trap R1R2
Drug: oxaliplatin — 85 mg/m2 IV infused over 2 hours
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin — 200 mg/m2 (Or levoleucovorin 100 mg/m2. If leucovorin is not available due to drug shortages the regimen should be administered with the leucovorin omitted) IV over 2 hours. Alternatively, leucovorin may be administered (via separate infusion lines) concurrently with oxaliplatin
  Other Names: CF; CFR; LV
Drug: fluorouracil — 400 mg/m2 IV bolus over 5-15 minutes, then 2400 mg/m2 continuous IV infusion over 46 hours.
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: Correlative Studies — Patients are required to have tissue available before enrolling on the study. A fresh biopsy is only required if there is insufficient material for analysis. Repeat tumor biopsies after 8 weeks of therapy are optional and will only be performed at the Ohio State University Medical Center.
  Other Names: laboratory biomarker analysis
Procedure: DCE MRI — Images at weeks 0, and after 8 weeks +/- 1 week of treatment (after Cycle 2).
  Other Names: Dynamic contrast-enhanced magnetic resonance imaging
Radiation: f18FDG-PET — 18FDG-PET is a functional imaging technique that relies on tumor uptake of radiolabeled tracer 18 fluorodeoxyglucose (18FDG). FDG-PET is a widely-used imaging modality in the detection and monitoring of a variety of metastatic cancers, including colorectal cancer (99-102).
  Other Names: 18FDG; FDG; fludeoxyglucose; F 18
Procedure: PET (positron emission tomography) — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
This phase II trial studies how well giving aflibercept together with combination chemotherapy works in treating patients with previously untreated colon or rectal cancer that is metastatic or locally advanced and cannot be removed by surgery. Aflibercept may stop the growth of colon or rectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving aflibercept together with combination chemotherapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression free survival (PFS) of patients with untreated metastatic colorectal cancer (mCRC) receiving the combination of modified leucovorin calcium, fluorouracil, oxaliplatin (FOLFOX6) (mFOLFOX6) and aflibercept.

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate (complete response [CR] + partial response [PR]) and the disease control rate (CR + PR + stable disease [SD]), as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, of patients with untreated mCRC receiving the combination of mFOLFOX6 and aflibercept.

II. To evaluate overall survival of patients with untreated mCRC receiving the combination of mFOLFOX6 and aflibercept.

III. To further characterize the safety and toxicity of the combination of mFOLFOX6 and aflibercept, including 60 day all-cause mortality.

IV. To describe patients with mCRC whose disease is rendered resectable as a consequence of therapy with the combination of mFOLFOX 6 and aflibercept.

TERTIARY OBJECTIVES:

I. To assess the use of dynamic imaging modalities including dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) and fluorodeoxyglucose (FDG)-positron emission tomography (PET) to evaluate changes in vascular permeability and FDG avidity and correlate with clinical efficacy (PFS, overall survival [OS], and response by RECIST 1.1).

II. To evaluate circulating levels of vascular endothelial growth factor A (VEGFA), phosphatidylinositol glycan anchor biosynthesis, class F (PlGF), soluble vascular endothelial growth factor receptor 2 (VEGF-R2), chemokine (C-X-C motif) ligand 12 (CXCL12) and chemokine (C-X-C motif) receptor 4 (CXCR4) as potential biomarkers for efficacy of aflibercept.

III. To evaluate for the presence of VEGF single nucleotide polymorphisms (SNPs) and whether any SNP(s), when detected, may be predictive of efficacy and/or toxicity of aflibercept.

IV. To assess microvessel density/tumor blood flow, capillary permeability and vessel normalization by tumor biopsy pre and post treatment with aflibercept.

V. To evaluate the presence of hypertension as a predictive biomarker for clinical efficacy of aflibercept.

OUTLINE:

Patients receive aflibercept intravenously (IV) over 1 hour followed by oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5-15 minutes and then continuously over 46 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of colorectal origin that is metastatic or locally advanced and unresectable
* Measurable disease, as defined by RECIST 1.1 criteria: one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with spiral computed tomography (CT) scan (CT scan slice thickness no greater than 5 mm) malignant lymph nodes will be considered measurable if they are >= 15 mm in short axis
* Must not have received any prior systemic therapy for metastatic or locally advanced CRC; prior VEGF inhibitors are not allowed
* Prior adjuvant therapy for CRC including fluoropyrimidines either alone or in combination with oxaliplatin is allowed, provided that all therapy was completed >= 12 months from cancer recurrence, therapy duration was =< 6 months, and all prior toxicities have completely resolved (residual grade 1 neuropathy is allowed)
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hemoglobin >= 9 g/dL (blood transfusion permitted to attain this value)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (may be =< 5x ULN if increase is due to metastatic disease)
* Creatinine =< 1.5 x institutional ULN or creatinine clearance >= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional U
* Urine protein:creatinine ratio (UPCR) < 1 or < 500 mg protein/24 hr
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* May not be receiving any other investigational agents
* Patients who have received any prior locoregional therapy for metastatic disease (e.g. radiofrequency/microwave ablation, Yttrium-90 radioembolization, transarterial chemoembolization, or surgical resection) are excluded
* Patients with known or suspected brain metastases, carcinomatous meningitis, uncontrolled seizure disorder, active intracranial bleeding or active neurologic disorder are excluded
* Patients with an active second primary malignancy or history of malignancy within the 5 years of enrollment are excluded, with the exception of non-melanoma skin cancers and cervical cancer which has been treated with curative therapy
* Grade >= 2 sensory neuropathy at the time of enrollment
* Major surgery within 4 weeks of study start date; the surgical incision should be fully healed prior to initiation of aflibercept
* Female or male patients of reproductive capacity unwilling to use methods appropriate to prevent pregnancy are excluded; effective contraception is required for at least 3 months following the last administration of aflibercept
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension (blood pressure [BP] must be well controlled < 160/90), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, or any condition that the principal investigator (PI) feels would make the patient ineligible
* Positive pregnancy screening test with a minimum sensitivity of 25 IU/L of human chorionic gonadotropin (hCG) within 72 hours of registration; breastfeeding women are also excluded
* History of pulmonary embolus within 3 months or deep venous thrombosis (DVT) within 4 weeks of enrollment; patients on anticoagulation must be on a stable dose of warfarin with a therapeutic-range international normalized ratio (INR) or on a stable dose of low molecular weight heparin
* Active congestive heart failure (New York Heart Association [NYHA] class II-IV)
* History of an arterial thrombotic vascular event including cerebrovascular accident (CVA), myocardial infarction (MI), unstable angina, coronary or peripheral arterial bypass graft, or transient ischemic attack (TIA) within 6 months
* Serious or non-healing wound, ulcer or bone fracture at the time of medication administration
* History of treatment-resistant peptic ulcer disease, erosive esophagitis, gastritis, or diverticulitis within 3 months
* History of gastrointestinal (GI) perforation within 5 years; current or prior intestinal fistulas are also excluded
* Known chronic infectious disease including human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS)
* History of major hemorrhage including gastrointestinal bleeding (grade 2-4), pulmonary hemorrhage, or clinically significant hemoptysis (> 1 tsp in 24 hours) within the last 5 years; patients with underling conditions that predispose to bleeding, such as bleeding diathesis, known esophageal varices, or tumor involving major vessels, are also excluded
* Inability to understand or comply with study protocol
* Known hypersensitivity to Chinese hamster ovary cell products or to recombinant human or murine antibodies, or any of the treatments in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hays, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (6):
- United States (6):
  - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aflibercept (Combination Chemotherapy)
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Aflibercept (Combination Chemotherapy): Patients receive aflibercept and fluorouracil and then continuously over 46 hours on days 1 and 15.If leucovorin is not available due to drug shortages the regimen should be administered with the leucovorin omitted. Correlative Studies are required to be available before enrolling on the study. A fresh biopsy is only required if there is insufficient material for analysis. Repeat tumor biopsies after 8 weeks of therapy are optional and will only be performed at the Ohio State University Medical Center.DCE MRI (dynamic contrast-enhanced magnetic resonance imaging)images at weeks 0, and after 8 weeks +/- 1 week of treatment(after Cycle 2). 18FDG-PET is a functional imaging technique that relies on tumor uptake of radiolabeled tracer 18 fluorodeoxyglucose (18FDG).FDG-PET is a widely-used imaging modality in the detection and monitoring of a variety of metastatic cancers,including colorectal cancer (99-102).
  aflibercept: 4 mg/kg as a 1-hour IV(intervenous) infusion oxaliplatin: 85 mg/m2 IV infused over 2 hours leucovorin: 200 mg/m2 (Or levoleucovorin 100 mg/m2. If leucovorin is not available due to drug shortages the regimen should be administered with the leucovorin omitted) IV over 2 hours. Alternatively, leucovorin may be administered (via separate infusion lines) concurrently with oxaliplatin fluorouracil: 400 mg/m2 IV bolus over 5-15 minutes, then 2400 mg/m2 continuous IV infusion over 46 hours.
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 56.9 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 43
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Progression-free at 15 Months
Description: Assuming that the number of treatment successes (alive and progression-free) is binomially distributed, proportion estimates along with their corresponding exact 95% confidence intervals will be calculated.
Time Frame: At 15 months from initiation of therapy
Measure: Number; unit: proportion of participants
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
proportion of participants | .482

2. Secondary Outcome: Objective Response Rate (ORR) Defined as the Proportion of Patients Who Achieve a PR or CR Based on RECIST 1.1 Criteria Divided by the Total Number of Evaluable Patients
Description: Summarized as a proportion with corresponding 95% confidence interval.
Time Frame: Up to 4 weeks post-treatment
Measure: Number; unit: proportion of participants
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
proportion of participants | 0.446

3. Secondary Outcome: Percentage of Patients Able to Undergo Surgery
Description: Summarized as a proportion with corresponding 95% confidence interval.
Time Frame: Up to 4 weeks post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
percentage of participants | 5.36

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Will be evaluated using the methods of Kaplan and Meier.
Time Frame: From study entry to the time of progressive disease and/or death, assessed up to 4 weeks post-treatment, assessed up to 4 years and 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
months | 7.82 [7.36 to 10.71]

5. Secondary Outcome: Overall Survival
Description: Will be evaluated using the methods of Kaplan and Meier.
Time Frame: From study entry to time of death due to any cause, assessed up to 4 weeks post-treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
months | 19.68 [16.23 to 25.79]

6. Secondary Outcome: Incidence of Severe (Grade 3+) Adverse Events or Toxicities, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Time Frame: Up to 4 weeks post-treatment
Measure: Number; unit: percentage of patients
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
percentage of patients
  Hypertension | 33.9
  Neutropenia | 25
  Thromboembolic events | 12.5
  Hypertriglyceridemia | 10.7

7. Secondary Outcome: Tolerability in Terms of Number of Patients Who Require Dose Modifications and/or Dose Delays
Time Frame: Up to 4 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
Participants | 50

8. Secondary Outcome: Proportion of Patients Who go Off Treatment Due to Adverse Reactions or Even Those Who Refuse Further Treatment for Lesser Toxicities That Inhibit Their Willingness to Continue Participation on the Trial
Time Frame: Up to 4 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept (Combination Chemotherapy)
Number analyzed (Participants) | 56
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected and graded for patients from start of study until study completion up to an average of 4 years.
Arm/Group | Aflibercept (Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/56
Serious Adverse Events (participants affected / at risk) | 7/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (Combination Chemotherapy) (N=56)
Hypertension (Vascular disorders) | 4 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 7 (7)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ileal obststruction (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (Combination Chemotherapy) (N=56)
Abdominal pain (Gastrointestinal disorders) | 11 (11)
Alanine aminotransferase increased (Investigations) | 15 (15)
Alkaline phosphatase increased (Investigations) | 24 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 31 (31)
Anorexia (Metabolism and nutrition disorders) | 18 (18)
Anxiety (Psychiatric disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 25 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Blood bilirubin increased (Investigations) | 8 (8)
Blurred vision (Eye disorders) | 6 (6)
Chills (General disorders) | 4 (4)
Cholesterol high (Investigations) | 21 (21)
Constipation (Gastrointestinal disorders) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine increased (Renal and urinary disorders) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 31 (31)
Dizziness (Nervous system disorders) | 16 (16)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Gastrointestinal disorders) | 17 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Fatigue (General disorders) | 34 (34)
Fever (General disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
Headache (Nervous system disorders) | 16 (16)
Hematuria (Renal and urinary disorders) | 10 (10)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (23)
Hyperkalemia (Investigations) | 7 (7)
Hypernatremia (Metabolism and nutrition disorders) | 5 (5)
Hypertension (Vascular disorders) | 37 (37)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 22 (22)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (20)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 10 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 13 (13)
Hypotension (Vascular disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5)
Lymphocyte count decreased (Investigations) | 22 (22)
Mucositis oral (Gastrointestinal disorders) | 31 (31)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 40 (40)
Cold Sensitivity (Nervous system disorders) | 4 (4)
Neutrophil count decreased (Investigations) | 28 (28)
Non cardiac chest pain (General disorders) | 6 (6)
Oral pain (Gastrointestinal disorders) | 5 (5)
Pain (General disorders) | 10 (10)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 (13)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (19)
Paresthesia (Nervous system disorders) | 14 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (33)
Platelet count decreased (Investigations) | 29 (29)
Proteinuria (Renal and urinary disorders) | 21 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 7 (7)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 5 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 11 (11)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 (10)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Thromboembolic event (Vascular disorders) | 11 (11)
Tremor (Nervous system disorders) | 4 (4)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (8)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 30 (30)
Weight loss (Investigations) | 16 (16)
White blood cell decreased (Investigations) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT01652196/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT01652196/ICF_001.pdf